CLINICAL TRIAL: NCT06927765
Title: Effect of Intraperitoneal Drain Placement on Postoperative Outcomes Following Laparoscopic Appendectomy in Adult Patients With Perforated Appendicitis: A Prospective, Multicenter, Randomized Controlled Trial
Brief Title: Effect of Intraperitoneal Drain Placement on Postoperative Outcomes Following Laparoscopic Appendectomy in Adult Patients With Perforated Appendicitis
Acronym: LADPA
Status: Active, not recruiting | Type: Observational
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Other Study IDs: LADPA
Record Dates: First submitted 2024-12-23; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Perforated Appendicitis
Keywords: Perforated appendicitis; abdominal drainage
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Biospecimen Retention: Samples Without DNA — Excision of the appendix Intraperitoneal pus
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Place an abdominal drain: Place an abdominal drain
  Interventions: Other: No abdominal drain is placed

INTERVENTIONS:
Other: No abdominal drain is placed — No abdominal drain is placed

SUMMARY:
Acute appendicitis is the most common acute abdomen, and a small number of patients can progress to perforated appendicitis, which has significantly higher complications than non-perforated appendicitis. Appendectomy is the only option for treating perforated appendicitis. Optimizing the diagnosis and treatment of perforated appendicitis is of great significance to improve its clinical outcomes and save medical resources.

There is a consensus that drainage should not be placed after surgery for non-perforated appendicitis, but the decision to place drainage for perforated appendicitis remains controversial. Several retrospective studies have shown no benefit in postoperative recovery and hospital stay, and may lead to increased infectious complications and longer hospital stays. A small number of prospective studies have shown similar conclusions, but the sample size is too small, most of them are children, and there is a lack of large-scale multicenter studies. The investigators' preliminary retrospective survey suggests that in China, most surgeons still commonly place drains for peace of mind after surgery with perforated appendicitis in adults without seeing a clear benefit, so there is a need for a multicenter prospective randomized controlled study to evaluate the need for drainage placement after perforated appendicitis and to guide clinical practice with evidence.

To study the effect of abdominal drainage on the postoperative clinical outcomes of adult patients with perforated appendicitis, mainly including: infectious complications (residual infection or abscess in the abdominal cavity, incision infection, fecal fistula, etc.), case fatality rate, pain score, length of hospital stay (LOS), quality of life (QOL) score, etc.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 years old (no upper limit);
* Perforated appendicitis or suspected perforated appendicitis who intends to undergo laparoscopic appendectomy;
* Patients and their families (or legal representatives) are able to understand the study protocol and voluntarily participate in this study, and sign informed consent.

Exclusion Criteria:

* Whole abdominal pus was found during the operation;
* Open or laparoscopic conversion to open appendectomy;
* Appendiceal tumors (including postoperative pathology)
* Pregnancy or perinatal period;
* AIDS, tuberculosis, liver cirrhosis, uremia, aplastic anemia, essential thrombocytopenia, inflammatory bowel disease, organ transplantation;
* Long-term or preoperative use of immunosuppressants/glucocorticoids/tumor chemotherapy drugs/targeted drugs/immunodrugs;
* Malignant tumors (including leukemia and lymphoma) disease status, recurrence/metastasis, and perioperative period;
* Drunk, drug abuse/drug addicts;
* Organ dysfunction/failure;
* Those who are transferred to the ICU for various reasons;
* Other conditions that the investigator considers unsuitable for inclusion (e.g., hyperthyroidism, bone marrow dysproliferative syndrome, acute myocardial infarction, acute cerebral infarction, diabetic ketoacidosis, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute perforated appendicitis >18 years of age
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Incision infection rate | From enrollment to 30 days postoperatively
  Superficial tissue infections, such as those at the site of the surgical Trocar foramen (epidermal or subcutaneous), do not enter the abdominal cavity
Incidence of intra-abdominal abscess | From enrollment to 30 days postoperatively
  Residual infection in the abdominal cavity forms an abscess.The incidence of intra-abdominal abscess after surgery will be compared between the two groups
Incidence of fecal leakage | From enrollment to 30 days postoperatively
  Dehiscence of the stump of the appendix causes fecal residue to enter the abdominal cavity

SECONDARY OUTCOMES:
Length of hospital stay | From enrollment to 30 days postoperatively
  Length of hospital stay（days，d）
Pain scores | From enrollment to 30 days postoperatively
  Visual Analog Score for pain
Quality of life scores | From enrollment to 30 days postoperatively
  The MOS item short from health survey, SF-36

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No
secrecy